CLINICAL TRIAL: NCT01567917
Title: Incidence of Venous Thromboembolism Following Surgery in Korean Patients With Colorectal Cancer; a Prospective Study
Brief Title: Incidence of Venous Thromboembolism Following Surgery in Patients With Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Keun-Wook Lee, Principal investigator, Seoul National University Bundang Hospital
Other Study IDs: CRC-SNUBH-2012-01
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Symptomatic Venous Thromboembolism; Asymptomatic Venous Thromboembolism
Keywords: Venous thromboembolism; Colorectal cancer; Postoperative period; detected on 5th~14th days after surgery (by doppler US) or the follow-up period of postoperative 1 month
MeSH Terms: conditions — Venous Thromboembolism; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Patients who gave a permission to this study and underwent doppler US (Doppler US cohort
  - Expected subject no.: 400 patients
  Interventions: Procedure: CRC surgery
- Group B: Patient who gave a permission to this study, but who did not receive doppler US (Although this group of patients did not undergo doppler US, these patients will be included as group B [simple observation cohort without doppler US examination])
  - Expected subject no.: 200 patients
  Interventions: Procedure: CRC surgery

INTERVENTIONS:
Procedure: CRC surgery — Patients will receive surgery for the treatment of CRC as routine clinical practice. These patients will be prospectively observed for the development of VTE(Group A; Doppler US cohort vs. Group B; Simple observation cohort)
  - Doppler US is not an intervention. The Doppler US is a non-invasive test (ultrasonography) for the detection of VTE

SUMMARY:
Venous thromboembolism (VTE) has harmful effects on morbidity and mortality of cancer patients. In Western VTE guidelines, all solid cancer patients receiving abdominal major surgery are strongly recommended to receive pharmacologic prophylactic anticoagulation such as low molecular weight heparin (LMWH) in the perioperative periods. These recommendations are based on the high incidence of postoperative VTE development in Western cancer patients. However, there have been many cumulative data about the effect of different ethnicity on the VTE development and more and more investigators and clinicians admit that Asian ethnicity has lower incidence of VTE than Western ethnicity. Therefore, it may not be advisable to apply Western guidelines as it is to the clinical situation of Asian cancer patients.

Although colorectal cancer (CRC) is one of the common cancers and the incidence is rapidly increasing in Asia, there have been few prospective data on the incidence of VTE development during the postoperative period in Asian CRC patients. To our knowledge, there have been a few small-sized prospective studies in Asia and thus clear conclusions could have not been drawn based on those studies. Most Korean colorectal surgeons think that the incidence of postoperative VTE development is very rare based on their own clinical experiences. They also have much concern about the complications such as bleeding that might be caused by routine use of pharmacologic thromboprophylaxis during the perioperative periods. Therefore, in most clinical situation, many Korean colorectal surgeons do not perform perioperative pharmacologic thromboprophylaxis using LMHW. Considering these clinical situations in Asia including Korea, the uncritical acceptance of Western guidelines may be inappropriate. The necessity of pharmacologic thrombo-prophylaxis can be answered only from our own prospective study on the incidence of postoperative VTE development after CRC surgery. Moreover, current surgical trend in cancer patients is minimally invasive approach such as laparoscopic surgery. However, the necessity of pharmacologic thromboprophylaxis in patients receiving laparoscopic cancer surgery has not been evaluated even in Western countries. Western guidelines also cannot exactly answer whether pharmacologic thromboprophylaxis is really necessary in cancer patients receiving laparoscopic cancer surgery. On above backgrounds, this study was designed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of colon or rectum
* Age ≥ 20 years
* Patients receiving curative or palliative abdominal surgery (lasting ≥ 30 minutes) (both open and laparoscopic surgery will be included)

Exclusion Criteria:

* No histological confirmation
* Patients who already have VTE (or pulmonary embolism) at the screening periods of this study
* Past medical history of VTE or pulmonary embolism
* Patients with the history of other cancer (Patients who were disease-free for > 5 years from previous other cancer is allowed to be included in this study)
* Patients with thrombophilia or other comorbidities requiring anticoagulation (i.e. atrial fibrillation or cerebral infarct requiring anticoagulation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CRC receiving curative or palliative surgery
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of symptomatic or asymptomatic VTE | 5~14 days after CRC surgery (by doppler venous ultrasound [US]) or the follow-up period of postoperative 1 month
  To evaluate the incidence of symptomatic or asymptomatic VTE detected by Doppler US during postoperative periods in patients with CRC receiving surgery

SECONDARY OUTCOMES:
Risk factors for the development of VTE | 5~14 days after CRC surgery (by doppler US) or the follow-up period of postoperative 1 month
  To identify risk factors for the development of VTE in this population

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea